CLINICAL TRIAL: NCT06862583
Title: Nordic Multicenter Study of Risk Factors, Surgical Treatment and Outcomes in Acute Type a Aortic Dissection
Brief Title: Nordic Consortium for Acute Type a Aortic Dissection-2
Acronym: NORCAAD-2
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Haukeland University Hospital (Other); Rigshospitalet, Denmark (Other); Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Leiden University Medical Center (Other); Skane University Hospital (Other); Odense University Hospital (Other); Oslo University Hospital (Other); Landspitali University Hospital (Other); Norrlands University Hospital (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Trondheim University Hospital (Other); University Hospital, Linkoeping (Other); Vastra Gotaland Region (Other Government); Uppsala University Hospital (Other); Blekinge County Council Hospital (Other); Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Christian Olsson, Associate professor, Karolinska Institutet
Other Study IDs: 2019-02087
Record Dates: First submitted 2025-01-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Aortic Dissection
Keywords: Open surgery; Risk factors; Outcomes; Mortality; Circulatory arrest; cerebral protection; bicuspid aortic valve
MeSH Terms: conditions — Aortic Dissection; Bicuspid Aortic Valve Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: surgery — Open heart surgery
Procedure: endovascular intervention — Aortic endovascular intervention

SUMMARY:
The Nordic Consortium for Acute Type A Aortic Dissection-2 (NORCAAD-2) is a multicenter research collaboration involving up to 19 units in the Nordic countries and one in The Netherlands. All patients referred for this condition is included, to outline detailed preoperative characteristics and risk factors as well as, for those operated, data on the operative procedure, the postoperative course including major and minor complications and, as the primary interest, mortality in short- and long-term perspective. The need for further procedures on the aorta will also be studied.

Acute type A Aortic Dissection (ATAAD) is a vascular emergency with very high case-fatality rate. The condition is realtively infrequent, and single units can rarely amass sufficient number of patients during a reasonable time to analyse also unusual variants in background, presentation, and management. Randomized controlled trials are unlikely, and large multicenter databases are the best source of knowledge for the foreseeable future. Other such databases exist, but NORCAAD-2 is more focused (only ATAAD) and more detailed than many counterparts, with the ability to extract unique information.

NORCAAD-2 is the extension and expansion of the original NORCAAD project. NORCAAD-2 includes more centers, more patients, more data and utilizes a novel on-line common database designed for the purpose.

The ultimate goal is to identify novel risk markers to help inform decisions on pre-emptive surgery (before ATAAD occurs); to outline superior perioperative techniques and strategies to optimize outcomes both short- and long-term; and to analyze variables related to major complications, in an effort to further reduce their incidence.

DETAILED DESCRIPTION:
Research project plan

NORCAAD - Nordic Consortium for acute type A aortic dissection Nordic multicenter study of risk factors, surgical treatment and outcomes in acute type A aortic dissection

Background Acute type A aortic dissection (ATAAD) is a major vascular disaster. The overall incidence is quoted at 2-3/100.000/year but probably higher due to undiagnosed cases, and certainly higher in specific age (60-65 years and up) and risk groups (eg. connective tissue disease such as Marfan syndrome). At around 70%, case-fatality rate is on par with for example ruptured abdominal aortic aneurysm. The inciting pathogenic event is a disruption of the ascending aortic endothelium, a so-called entry tear (when located in the arch or descending aorta, the dissection is generally referred to as type B, and this form will not be further discussed). From this entry tear, shear stress of the bloodstream dissects the aortic wall layers, producing intense pain, but also a lethal threat with risk of rupture and tamponade, malperfusion of vital aortic branches, and aortic valve dysfunction with regurgitation and heart failure. Little, however, is known about risk factors. Hypertension is common in this patient group. Some cardiovascular abnormalities such as bicuspid aortic valve, aortic arch anomalies, or aortic coarctation are thought to increase risk, as is a pre-existing ascending aortic aneurysm or known cases of aortic dissection or aneurysm among first-degree relatives. Based on the poor prognosis, there is general consensus that ATAAD is treated surgically, with repair (graft replacement) of the ascending aorta. Data supports that this treatment is given as soon as possible, as mortality increase by the hour in ATAAD. Even with surgical therapy, early (30-day or in-hospital) mortality approaches 20% and severe complications (stroke, renal and respiratory insufficiency, multisystem organ failure) remain at substantial 10-20% prevalence each. Long-term outcomes for early survivors are acceptable, albeit not normal. Specifically, need for reintervention and reoperation due either to local or remote aortic conditions, persists or occur even long after primary surgery, necessitating often life-long surveillance.

Overview: knowledge gaps Despite a vast literature on ATAAD, many aspects remain poorly understood and/or controversial, and there are very few issues characterized by broad consensus. In parallel, treatment modalities evolve and successful concepts from elective aortic surgery is implemented also in the management of ATAAD and their respective roles remain to be determined.

Risk factors and predisposing conditions As mentioned, bicuspid aortic valve (BAV) is regarded as over-represented in ATAAD patients; its prevalence is estimated at 1-2% in a general population and often 5-15% in ATAAD case series. However, very little detail is known about what subtypes (according to the Sievers classification) are more common and if the are associated with pre-ATAAD dilatation of the aortic root and/or ascending aorta or with a valve dysfunction (and if so, more commonly stenosis or regurgitation?). It has been shown that ascending aortic diameter by itself is not a good predictor of ATAAD. Therefore, other radiological findings are explored to predict ATAAD risk. Aortic arch branching anomalies are one such feature, where specific aortic arch branch patterns seem prevalent. Such risk markers could be important in the decision-making process for prophylactic aortic surgery in selected patients.

Preoperative complications Currently, the primary differential diagnosis, i.e. acute coronary syndrome (ACS), poses a problem, since it mandates early and powerful antithrombotic and antiplatelet therapy, which in turn can be detrimental from a surgical point of view. Diagnosis of ACS is increasingly often made in the pre-hospital setting, in turn increasing the risk for misdiagnosis and -treatment. The exact magnitude of this problem is not known, nor is its net effect in surgical outcomes; survival, but also bleeding complications, transfusion requirements and need for hemostatic agents.

In general, malperfusion syndromes, i.e. end-organ ischemia caused by arterial compromise due to the dissection, are well-known to increase mortality and morbidity. Fortunately, some variants are infrequent, eg. coronary and intestinal malperfusion. Therefore, their optimal management is less well outlined. A subset will even be denied surgery, if deemed futile. It would be of importance, however, to always offer surgical treatment if it offers a potential survival benefit.

Surgical procedures Most common, and most conservative, is to replace the ascending aorta with a vascular prosthesis from above the coronary orifices to below the arch vessels. If addressing the potential lethal ATAAD complications (rupture, tamponade, aortic regurgitation, coronary or distal malperfusion) it is adequate, and confers lowest possible surgical risk. However, in several instances it may be insufficient, for example when aortic regurgitation is severe, the aortic root or arch dilated, or the intimal tear continues through the arch, or there is an underlying connective tissue disease heralding late complications with conservative approaches. Such instances may force more extensive and complex surgical procedures, with variants of aortic valve, root, and arch replacements or repairs. Over time, such procedures have been reported feasible, and with growing experience in elective settings, they are more often advocated as primary ATAAD procedures as well - to avoid possible late complications and reoperations.

Extracorporeal circulation Aspects of extracorporeal circulation (ECC) with the heart-lung machine include how to cannulate the arterial system in ATAAD and how to perform ECC, more specifically: hypothermic circulatory arrest (HCA) or not? If so, at what temperature; body (core) and brain? And aided by which form of cerebral perfusion? Numerous techniques are reported with often similar, but sometimes contradicting, outcomes. The basic principles of speed of establishing ECC, avoidance of ECC-induced malperfusion, and a minimization of embolic and hypofperfusion risk related to ECC are agreed upon, but not the appropriate measures to reach them.

Postoperative course A patient surviving ATAAD and ATAAD surgery remains at great risk of suffering severe complications, cf. above. What steps are needed to prevent and treat such complications needs to be further explored, since they are common, and since late survival may be satisfying, if the index hospital period is managed. A greater understanding is needed to adequately prognose, inform patients and relatives, and allocated health care resources. For example, is embolic stroke different from watershed stroke in these aspects? Which patients will recover renal function after acute renal injury, and to what extent? What factors contribute to critical illness polymyopathy/neuropathy and how does it affect late outcomes?

Late outcomes What (mainly surgical) factors contribute to late reoperation? In an early (pseudoaneurysm, root dilatation, aortic regurgitation) and late (aneurysm formation)? How long does these conditions need to occur? How does endovascular repair techniques affect outcomes of secondary procedure? These and similar questions are of utmost importance to the survivors of ATAAD, since a significant proportion of them might end up there.

This brief summary also serves as examples of the research issues addressed by NORCAAD. Each of the listed knowledge gaps will be investigated as separate substudies; each with study hypotheses to test or explicit research questions to be answered.

Conditions for ATAAD clinical research ATAAD will, reasonably, never be the subject of a randomized controlled trial. Allocation to surgical treatment or not is impossible. Allocation to different surgical procedures is impossible. Allocation to different modes of ECC is impossible. Minor details, such as use of different pharmacological agents, could be possible and has even been studied, but without impact on management. Many patients would never be able to give informed consent, they are in too much pain, they are to mentally obtunded, unconscious or, more often, need to be rushed to surgery without unnecessary, let alone potentially dangerous, delay. In this sense, ATAAD practice will never be truly evidence-based [8]. Single center case series are affluent. Outcomes of specific surgical procedures, ECC regimens, or other management aspects are reported; increasingly often with very good results almost thought impossible only a decade ago. But they lack sizeable study populations, adequate control groups and, above all, generalizability since they are often based on site-specific unique conditions such as around-the-clock aortic teams, hybrid OR suites, home-made vascular and endovascular devices. In addition, publication bias will remain, with negative outcomes less frequently reported. Large study populations accrued during as short and recent time-frame as possible (to truly reflect current practices) in "real world" conditions and with meticulous follow-up would serve the best possible base. Multicenter studies performed in a comparably homogenous population and health care-system would be the best option. NORCAAD is exactly that [9].

NORCAAD

NORCAAD is an acronym for Nordic Consortium for acute type A aortic dissection. The purpose is to create a common, multicenter, multinational, contemporary and growing database with extended follow-up, to fill in the above listed, among others, knowledge gaps with as good clinical data as currently possible. NORCAAD will include 19 centers from all Nordic countries:

DENMARK Aarhus, Copenhagen, Odense FINLAND Helsinki, Kuopio, Tampere, Turku ICELAND Reykjavik NORWAY Bergen, Oslo, Trondheim SWEDEN Gothenburg, Karlskrona, Linköping, Lund, Stockholm, Umeå, Uppsala, Örebro AND, as an associate member, The Leiden University Medical Centre (LUMC) for a total of 20 participating centers.

An estimated 450 ATAAD cases (range 5-50 per unit) are performed annually, along with a (hitherto unknown) number of ATAAD surgical candidates managed non-operatively. Perioperative techniques remain at the discretion of the treating surgeons at each unit; together creating a representative view of current practice. A number of clinical and demographical variables, of which many notably are not available in other studies, are collected in a common, dedicated, on-line database. Database screenshots are shown below to illustrate.

NORCAAD aims to include all consecutive ATAAD patients presented to participating centers since January 1, 2000 and onwards. No exclusion criteria will be applied other than age >18 years (which in practice is exceedingly rare). Demographical, clinical, examination, intra- and postoperative as well as follow-up and survival status data will be collected for at least 2500 patients and, at the termination of inclusion, up to 5000 patients, making NORCAAD on of the worlds' largest multinational multicenter ATAAD databases.

Statistical methods Variable types include continuous, dichotomous, categorical, and ordinal data, as well as dates for analyses of time-related events. Standard statistical methods are employed for analysis, including bivariate and multivariable analysis using logistic regression. Group comparisons are made using parametric and non-parametric tests as suitable, based on individually specified study hypotheses. Time-dependent analyses employ Kaplan-Meier methods for estimation of survival, log-rank tests for group comparisons, and Cox proportional hazards analysis for hazard ratios. Competing risks are accounted for when applicable. Further data exploration using for example propensity score methods are used when adequate. Statistical analyses are performed in collaboration with biostatisticians.

Clinical implications

* Improved characterization of prognostic factors will contribute to improved selection of surgical candidates and identify non-candidates with increased accuracy; of importance to ATAAD sufferers, their relatives, and to health care resource allocation.
* Identification of non-diameter based imaging criteria (BAV subtype, arch anomalies) may alter indications for prophylactic aortic surgery, with dramatically reduced risks.
* Detailed evaluation of merits of different intraoperative procedures in short and long-term perspective is essential to understand when different surgical solutions are indicated, with an ultimate goal of individualized treatment to optimize outcomes.
* Characterization of specific very-high risk patient groups may contribute to regionalization of care, creation of aortic centers and similar health care system adaptations
* True long-term follow-up is needed to detect long-term outcomes: survival but also intercurrent morbidity and need for reinterventions, endovascular or open surgical, in turn instrumental to decide on surveillance length and intervals.

To summarize, NORCCAD data and findings may in several ways have significant impact on many crucial aspects of ATAAD management and move it towards practice based on solid clinical data. Current guidelines, North American and European, will be updated and NORCAAD aims to provide new data to improve those guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Acute (within 14 days of onset) type A aortic dissection or similar acute aortic syndrome

Exclusion Criteria:

* Age <18 years at onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute type A aortic dissection referred to any of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Early mortality | 30 days
  Mortality within 30 days of referral or operation

SECONDARY OUTCOMES:
Late mortality | >30 days
  Mortality late after referral or operation
Reintervention | throughout study period
  Any reintervention (endovascular, open surgical) on the aorta

OTHER OUTCOMES:
Permanent neurological damage | 30 days
  Stroke or spinal cord infarction with permament neurological symptoms
Temporary neurological damage | 30 days
  Transitory ischemic attack, minor stroke, coma or unconsciousness, confusion or other new neurological symptoms resolving before discharge
Renal insufficiency | 30 days
  Renal insufficiency (as graded and described by various classification systems)
Re-exploration | 72 hours
  Re-exploration for control of bleeding or tamponade

CONTACTS AND LOCATIONS:
Overall Officials: Christian Olsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eleid MF, Forde I, Edwards WD, Maleszewski JJ, Suri RM, Schaff HV, Enriquez-Sarano M, Michelena HI. Type A aortic dissection in patients with bicuspid aortic valves: clinical and pathological comparison with tricuspid aortic valves. Heart. 2013 Nov;99(22):1668-74. doi: 10.1136/heartjnl-2013-304606. Epub 2013 Sep 4. PMID 24006455
- [Background] Myrmel T, Lai DT, Miller DC. Can the principles of evidence-based medicine be applied to the treatment of aortic dissections? Eur J Cardiothorac Surg. 2004 Feb;25(2):236-42; discussion 242-5. doi: 10.1016/j.ejcts.2003.11.022. PMID 14747119
- [Background] Geirsson A, Ahlsson A, Franco-Cereceda A, Fuglsang S, Gunn J, Hansson EC, Hjortdal V, Jarvela K, Jeppsson A, Mennander A, Nozohoor S, Olsson C, Wickbom A, Zindovic I, Gudbjartsson T. The Nordic Consortium for Acute type A Aortic Dissection (NORCAAD): objectives and design. Scand Cardiovasc J. 2016 Oct-Dec;50(5-6):334-340. doi: 10.1080/14017431.2016.1235284. Epub 2016 Sep 26. PMID 27615395
- [Background] Hiratzka LF, Bakris GL, Beckman JA, Bersin RM, Carr VF, Casey DE Jr, Eagle KA, Hermann LK, Isselbacher EM, Kazerooni EA, Kouchoukos NT, Lytle BW, Milewicz DM, Reich DL, Sen S, Shinn JA, Svensson LG, Williams DM; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines; American Association for Thoracic Surgery; American College of Radiology; American Stroke Association; Society of Cardiovascular Anesthesiologists; Society for Cardiovascular Angiography and Interventions; Society of Interventional Radiology; Society of Thoracic Surgeons; Society for Vascular Medicine. 2010 ACCF/AHA/AATS/ACR/ASA/SCA/SCAI/SIR/STS/SVM Guidelines for the diagnosis and management of patients with thoracic aortic disease. A Report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, American Association for Thoracic Surgery, American College of Radiology,American Stroke Association, Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, Society of Interventional Radiology, Society of Thoracic Surgeons,and Society for Vascular Medicine. J Am Coll Cardiol. 2010 Apr 6;55(14):e27-e129. doi: 10.1016/j.jacc.2010.02.015. No abstract available. PMID 20359588
- [Background] Authors/Task Force Members; Czerny M, Grabenwoger M, Berger T, Aboyans V, Della Corte A, Chen EP, Desai ND, Dumfarth J, Elefteriades JA, Etz CD, Kim KM, Kreibich M, Lescan M, Di Marco L, Martens A, Mestres CA, Milojevic M, Nienaber CA, Piffaretti G, Preventza O, Quintana E, Rylski B, Schlett CL, Schoenhoff F, Trimarchi S, Tsagakis K; EACTS/STS Scientific Document Group; Siepe M, Estrera AL, Bavaria JE, Pacini D, Okita Y, Evangelista A, Harrington KB, Kachroo P, Hughes GC. EACTS/STS Guidelines for Diagnosing and Treating Acute and Chronic Syndromes of the Aortic Organ. Ann Thorac Surg. 2024 Jul;118(1):5-115. doi: 10.1016/j.athoracsur.2024.01.021. Epub 2024 Feb 26. No abstract available. PMID 38416090
- [Background] Mazzolai L, Teixido-Tura G, Lanzi S, Boc V, Bossone E, Brodmann M, Bura-Riviere A, De Backer J, Deglise S, Della Corte A, Heiss C, Kaluzna-Oleksy M, Kurpas D, McEniery CM, Mirault T, Pasquet AA, Pitcher A, Schaubroeck HAI, Schlager O, Sirnes PA, Sprynger MG, Stabile E, Steinbach F, Thielmann M, van Kimmenade RRJ, Venermo M, Rodriguez-Palomares JF; ESC Scientific Document Group. 2024 ESC Guidelines for the management of peripheral arterial and aortic diseases. Eur Heart J. 2024 Sep 29;45(36):3538-3700. doi: 10.1093/eurheartj/ehae179. No abstract available. PMID 39210722
- [Background] Girdauskas E, Disha K, Borger MA, Kuntze T. Risk of proximal aortic dissection in patients with bicuspid aortic valve: how to address this controversy? Interact Cardiovasc Thorac Surg. 2014 Mar;18(3):355-9. doi: 10.1093/icvts/ivt518. Epub 2013 Dec 12. PMID 24336701
- [Background] Conzelmann LO, Weigang E, Mehlhorn U, Abugameh A, Hoffmann I, Blettner M, Etz CD, Czerny M, Vahl CF; GERAADA Investigators. Mortality in patients with acute aortic dissection type A: analysis of pre- and intraoperative risk factors from the German Registry for Acute Aortic Dissection Type A (GERAADA). Eur J Cardiothorac Surg. 2016 Feb;49(2):e44-52. doi: 10.1093/ejcts/ezv356. Epub 2015 Oct 28. PMID 26510701
- [Background] Evangelista A, Isselbacher EM, Bossone E, Gleason TG, Eusanio MD, Sechtem U, Ehrlich MP, Trimarchi S, Braverman AC, Myrmel T, Harris KM, Hutchinson S, O'Gara P, Suzuki T, Nienaber CA, Eagle KA; IRAD Investigators. Insights From the International Registry of Acute Aortic Dissection: A 20-Year Experience of Collaborative Clinical Research. Circulation. 2018 Apr 24;137(17):1846-1860. doi: 10.1161/CIRCULATIONAHA.117.031264. PMID 29685932
- [Background] Howard DP, Banerjee A, Fairhead JF, Perkins J, Silver LE, Rothwell PM; Oxford Vascular Study. Population-based study of incidence and outcome of acute aortic dissection and premorbid risk factor control: 10-year results from the Oxford Vascular Study. Circulation. 2013 May 21;127(20):2031-7. doi: 10.1161/CIRCULATIONAHA.112.000483. Epub 2013 Apr 18. PMID 23599348
- [Background] Olsson C, Thelin S, Stahle E, Ekbom A, Granath F. Thoracic aortic aneurysm and dissection: increasing prevalence and improved outcomes reported in a nationwide population-based study of more than 14,000 cases from 1987 to 2002. Circulation. 2006 Dec 12;114(24):2611-8. doi: 10.1161/CIRCULATIONAHA.106.630400. Epub 2006 Dec 4. PMID 17145990
- [Background] Melvinsdottir IH, Lund SH, Agnarsson BA, Sigvaldason K, Gudbjartsson T, Geirsson A. The incidence and mortality of acute thoracic aortic dissection: results from a whole nation study. Eur J Cardiothorac Surg. 2016 Dec;50(6):1111-1117. doi: 10.1093/ejcts/ezw235. Epub 2016 Jun 22. PMID 27334108